CLINICAL TRIAL: NCT05124938
Title: Assessment of CA19-9 in Patients' With Thyroid Malignancies
Brief Title: Assessment of CA 19-9 in Patients' With Thyroid Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Ashraf Ahmed, Resident of clinical and chemical pathology, Sohag University
Other Study IDs: Soh-Med-21-10-11
Record Dates: First submitted 2021-10-26; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Thyroid Cancer
Keywords: CA19-9
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Healthy individuals
  Interventions: Diagnostic Test: Laboratory investigations for control: a-Complete blood count. b-Liver function test. c-kidney function test. d-thyroid-stimulating hormone,T3 and T4. e-Assessment of levels of CA19-9.
- Group 2: patients with localized thyroid malignancy
  Interventions: Diagnostic Test: Laboratory investigations for control: a-Complete blood count. b-Liver function test. c-kidney function test. d-thyroid-stimulating hormone,T3 and T4. e-Assessment of levels of CA19-9.
- Group 3: patients with metastatic thyroid malignancy
  Interventions: Diagnostic Test: Laboratory investigations for control: a-Complete blood count. b-Liver function test. c-kidney function test. d-thyroid-stimulating hormone,T3 and T4. e-Assessment of levels of CA19-9.

INTERVENTIONS:
Diagnostic Test: Laboratory investigations for control: a-Complete blood count. b-Liver function test. c-kidney function test. d-thyroid-stimulating hormone,T3 and T4. e-Assessment of levels of CA19-9. — a-Complete blood count. b-Liver function test. c-kidney function test d-thyroid-stimulating hormone,T3 and T4. e-Assessment of levels of CA19-9.

SUMMARY:
Thyroid cancer is a rare disease that represents approximately 3.8% of all new cancer cases.Incidence of thyroid cancer in north Africa about 2.8% of all new cancer cases with mortality rate about 0.73%.Thyroid malignancies are classified into different groups as follows:Papillary thyroid cancer which is the most common form of thyroid cancer form about 80-90% of all thyroid cancers,Follicular thyroid cancer that forms about 10-15% of all thyroid cancers,Anaplastic thyroid cancer that forms less than 2% of all thyroid cancers,Medullary thyroid cancer that forms about 5-10% and other rare types include thyroid lymphoma, and thyroid sarcoma.

Medullary thyroid carcinoma (MTC) is a rare disease, and its classic tumor marker is calcitonin. However, recently, very aggressive cases have been reported to also secrete carbohydrate antigen 19-9 (CA19-9), and its role as a marker of worse prognosis has been questioned.

DETAILED DESCRIPTION:
Thyroid cancer is a rare disease that represents approximately 3.8% of all new cancer cases.Incidence of thyroid cancer in north Africa about 2.8% of all new cancer cases with mortality rate about 0.73%.Thyroid malignancies are classified into different groups as follows:Papillary thyroid cancer which is the most common form of thyroid cancer form about 80-90% of all thyroid cancers,Follicular thyroid cancer that forms about 10-15% of all thyroid cancers,Anaplastic thyroid cancer that forms less than 2% of all thyroid cancers,Medullary thyroid cancer that forms about 5-10% and other rare types include thyroid lymphoma, and thyroid sarcoma.

Medullary thyroid carcinoma (MTC) is a rare disease, and its classic tumor marker is calcitonin. However, recently, very aggressive cases have been reported to also secrete carbohydrate antigen 19-9 (CA19-9), and its role as a marker of worse prognosis has been questioned.

CA19-9 was originally described as a gastrointestinal system and pancreas specific tumor marker. Immunohistochemical studies have demonstrated that CA19-9 is expressed in both differentiated and anaplastic thyroid carcinomas. Increased serum levels of CA 19-9 were reported in few patients with anaplastic thyroid cancer.The idea that CA19.9 could be predictive of mortality in MTC stems from early research which showed that serum creatinine and increased carcinoembryonic antigen levels were not important markers in MTC, but that Ca19.9, which is secreted in MTC, was significantly associated with progressive disease.

ELIGIBILITY:
* Inclusion Criteria: Patients with malignant thyroid tumors.
* Exclusion criteria: Patients with benign thyroid tumors ,Patients not known to have pancreatic disease.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group1: age and sex matched healthy control individuals. Group2: patients with localized thyroid malignancy. Group3: patients with metastatic thyroid malignancy.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum levels of CA19-9 in patients' with thyroid malignancies. | within 3 days after collection of the samples
  Measurement of serum levels of CA19-9 in patients' with thyroid malignancies by chemiluminescence methods of study on I flash device.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ashraf, Principal Investigator — Sohag University
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No